CLINICAL TRIAL: NCT06491563
Title: A Phase 2 Multicenter, Open-label Study to Investigate the Efficacy and Safety of Regimens Containing BRII-179, BRII-835, and Pegylated Interferon Alpha (PEG-IFNα) for the Treatment of Chronic Hepatitis B Virus (HBV) Infection (ENRICH)
Brief Title: Study to Investigate the Efficacy and Safety of Regimens Containing BRII-179, BRII-835, and PEG-IFNα Treating Chronic Hepatitis B Virus (HBV) Infection (ENRICH)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brii Biosciences Limited (Industry)
Collaborators: Vir Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRII-179-835-002
Record Dates: First submitted 2024-06-28; First posted 2024-07-09 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: For Treatment of Chronic Hepatitis B Virus Infection

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BRII-179 (longer dose interval) followed by BRII-835 + PEG-IFNα (Experimental): Participants will receive BRII-179 of a longer dose interval, followed by BRII-835 and PEG-IFNα combination therapy.
  Interventions: Biological: BRII-179; Drug: BRII-835 (VIR-2218); Biological: PEG-IFNα
- BRII-179 (shorter dose interval) followed by BRII-835 + PEG-IFNα (Experimental): Participants will receive BRII-179 of a shorter dose interval, followed by BRII-835 and PEG-IFNα combination therapy.
  Interventions: Biological: BRII-179; Drug: BRII-835 (VIR-2218); Biological: PEG-IFNα

INTERVENTIONS:
Biological: BRII-179 — BRII-179 will be given via intramuscular injection
Drug: BRII-835 (VIR-2218) — BRII-835 will be given via subcutaneous injection
  Other Names: elebsiran
Biological: PEG-IFNα — PEG-IFNα will be given via subcutaneous injection
  Other Names: Pegylated interferon alfa

SUMMARY:
This study will evaluate the efficacy and safety of the regimens containing BRII-179, BRII-835, and PEG-IFNα in adult participants with chronic hepatitis B virus (HBV) infection receiving nucleos(t)ide reverse transcriptase inhibitors (NRTIs) as background therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female aged 18-60 years.
* 2. Body mass index ≥ 18 kg/m2 and ≤ 32 kg/m2.
* 3. Chronic HBV infection for ≥ 6 months.
* 4. On NRTI therapy for ≥ 6 months.

Exclusion Criteria:

* 1. Any clinically significant chronic or acute medical condition that makes the participant unsuitable for participation.
* 2. Significant liver fibrosis or cirrhosis.
* 3. History or evidence of drug or alcohol abuse.
* 4. History of intolerance to SC or IM injection.
* 5. History of chronic liver disease from any cause other than chronic HBV infection.
* 6. History of hepatic decompensation.
* 7. Contraindications to the use of PEG-IFNα.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants achieving HBsAg seroclearance at 24 weeks post end of study treatment in anti-HBs responders compared with non-responders defined at protocol-specific timepoint | 24 weeks post end of treatment

SECONDARY OUTCOMES:
Percentage of participants achieving HBsAg seroclearance at 24 weeks post end of study treatment in anti-HBs responders compared with non-responders defined at protocol-specific timepoint (in participants with lower baseline HBsAg levels) | 24 weeks post end of treatment
Percentage of participants with treatment-emergent adverse events (TEAEs) | 24 weeks post NRTI discontinuation
Percentage of participants with serious adverse events (SAEs) | 24 weeks post NRTI discontinuation
Percentage of participants with abnormalities in hematology, chemistry, and/or coagulation parameters | 24 weeks post NRTI discontinuation
Appearance of anti-HBs at any timepoint | 24 weeks post NRTI discontinuation
Titers of anti-HBs at any timepoint | 24 weeks post NRTI discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofei Chen, Study Director — Brii Biosciences Limited
Locations (12):
- China (12):
  - Investigative Site 86004, Beijing, Beijing Municipality
  - Investigative Site 86009, Beijing, Beijing Municipality
  - Investigative Site 86015, Xiamen, Fujian
  - Investigative Site 86012, Foshan, Guangdong
  - Investigative Site 86001, Guangzhou, Guangdong
  - Investigative Site 86013, Guangzhou, Guangdong
  - Investigative Site 86002, Shenzhen, Guangdong
  - Investigative Site 86003, Shanghai, Shanghai Municipality
  - Investigative Site 86008, Shanghai, Shanghai Municipality
  - Investigative Site 86007, Chengdu, Sichuan
  - Investigative Site 86011, Chengdu, Sichuan
  - Investigative Site 86005, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No